CLINICAL TRIAL: NCT03255239
Title: Randomized Clinical Trial Comparing Open Preperitoneal Mesh, Retromuscular Mesh and Suture Repair for Abdominal Wall Hernias Less Than 3 cm Diameter
Brief Title: Open Preperitoneal Mesh Versus Retromuscular Mesh Versus Suture Repair for Abdominal Wall Hernias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital Universitaire Taher Sfar (Other Government)
Responsible Party: Principal Investigator, Mohamed Ali Chaouch, Resident of general surgery, Hôpital Universitaire Taher Sfar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Abdominal wall hernia repair
Record Dates: First submitted 2017-08-15; First posted 2017-08-21 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Ventral Hernia; Ventral Incisional Hernia; Umbilical Hernia
Keywords: ventral hernia; Open mesh repair; Polyester mesh; Preperitoneal; Retromuscular
MeSH Terms: conditions — Hernia, Ventral; Hernia, Umbilical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preperitoneal mesh repair (Experimental): Ventral hernia repair using polyester preperitoneal mesh repair
  Interventions: Procedure: Ventral hernia repair
- Retromuscular mesh repair (Experimental): Ventral hernia repair using polyester retromuscular mesh repair
  Interventions: Procedure: Ventral hernia repair
- Suture repair (Experimental): Ventral hernia repair using suture repair
  Interventions: Procedure: Ventral hernia repair

INTERVENTIONS:
Procedure: Ventral hernia repair — Hernia repair is a surgical procedure to return an organ that protrudes through a weak area of muscle to its original position.
  Other Names: retromuscular mesh repair; preperitoneal mesh repair; suture hernia repair

SUMMARY:
Randomized clinical trial comparing open preperitoneal mesh, retromuscular mesh and suture repair for ventral hernias less than 3 cm diameter

DETAILED DESCRIPTION:
Many techniques of ventral hernias repair have been reported. It is shown that open mesh hernia repairs have low recurrence and low complication rates then suture repair. But for hernias less than 3 cm some surgeons defend the treatment by suture. The main variable of interest is the location of mesh placement compared to suture repair. The investigator will compare in a prospective randomized clinical trial three techniques of abdominal wall hernia repair: preperitoneal polyester mesh, retromuscular polyester mesh and suture for hernias less than 3 cm. All patients underwent general anesthesia. The investigators used Polyester-based mesh because it has shown minimal shrinkage and excellent tissue ingrowth in animal models. Operative notes were physician-abstracted and the presence, type, and location of mesh prosthesis was recorded. Independent variables of interest were patient-level demographics (age and sex), facility where hernia repair occurred, year of hernia repair, preoperative comorbid conditions, history of prior repair, and intraoperative variables. The results compared postoperative pain was evaluated using a visual analogue scale (range, 0-10) on the day of the first outpatient visit, operating time evaluated as skin-to-skin time, drain management and both of early and late complications including seroma and hematoma formation, wound infection, fistula formation and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Vebtral hernia or post incisional hernia diameter < 3 cm
* Male or female aged between 18 and 90 year-old
* Elective surgery for ventral hernia

Exclusion Criteria:

* Any contraindication to the prosthetic treatment.
* Any hernia or incisional hernia with a collar strictly greater than 3 cm.
* Previous hernia mesh repaired
* contraindication for general anaesthesia
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rates | One year
  Late complications of ventral hernia repair

SECONDARY OUTCOMES:
Operating time | 15 to 90 minutes
  operating time evaluated as skin-to-skin time
Early complication | 30 days
  Early complicaion including seroma and hematoma formation, wound infection and fistula
Postoperative pain | 6, 12 and 24 hours
  Postoperative pain evaluated using a visual analogue scale (range, 0-10) on the day of the first outpatient visit

CONTACTS AND LOCATIONS:
Locations (1):
- Taher Sfar Hospital, Mahdia, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided